CLINICAL TRIAL: NCT04615429
Title: Double-blind, Randomized, Controlled, Clinical Trial to Assess the Efficacy of Allogenic Mesenchymal Stromal Cells in Patients With Acute Respiratory Distress Syndrome Due to COVID-19
Brief Title: Clinical Trial to Assess the Efficacy of MSC in Patients With ARDS Due to COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cristina Avendaño Solá (Other)
Responsible Party: Sponsor-Investigator, Cristina Avendaño Solá, Head of Clinical Pharmacology Deptarment, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-AT; 2020-002193-27 (EudraCT Number)
Record Dates: First submitted 2020-10-25; First posted 2020-11-04 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19 Pneumonia
Keywords: Acute Respiratory Distress Syndrome; COVID-19 Pneumonia; Mesenchymal stromal cells; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stromal cells (Experimental): Approximately 1x10E6 MSC/kg
  Interventions: Biological: Mesenchymal stromal cells
- Control group (Placebo Comparator): Solution identical to experimental treatment, without the MSC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal stromal cells — Administration of one single dose of allogenic Mesenchymal stromal cells
  Arms: Mesenchymal Stromal cells
Other: Placebo — Administration of placebo (solution identical to experimental treatment, without the MSC)
  Arms: Control group

SUMMARY:
A double-blind, randomized, controlled, clinical trial to evaluate the efficacy and safety of MSC (mesenchymal stromal cells) intravenous administration in patients with COVID-induced ARDS compared to a control arm.

DETAILED DESCRIPTION:
A double-blind, randomized, controlled, clinical trial to evaluate the efficacy and safety of MSC (mesenchymal stromal cells) intravenous administration in patients with COVID-induced ARDS compared to a control arm.

All trial participants will receive SOC*.

Randomization will be 1:1 between:

* Treatment arm: allogenic MSC.
* Control arm: Placebo (solution with the same composition as the experimental treatment, without the MSC).

  * SOC can include any medicines that are being used in clinical practice (e.g. lopinavir/ritonavir; hydroxy/chloroquine, tocilizumab, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent prior to performing study procedures (witnessed oral consent with written consent by representatives will be accepted to avoid paper handling). Written consent by patient or representatives will be obtained whenever possible.
2. Adult patients ≥18 years of age at the time of enrolment.
3. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, in oropharyngeal swabs or any other relevant specimen obtained during the course of the disease. Alternative tests (e.g., rapid antigenic tests) are also acceptable as laboratory confirmation if their specificity has been accepted by the Sponsor.
4. Moderate to severe ARDS (PaO2/FiO2 ratio equal or less than 200 mmHg) for less than 96 hours at the time of randomization.
5. Patients requiring invasive ventilation are eligible within 72 hours from intubation.
6. Eligible for ICU admission, according to the clinical team.

Exclusion Criteria:

1. Imminent and unavoidable progression to death within 24 hours, irrespective of the provision of treatments (in the opinion of the clinical team).
2. "Do Not Attempt Resuscitation" order in place.
3. Any end-stage organ disease or condition, which in the investigator's opinion, makes the patient an unsuitable candidate for treatment.
4. History of a moderate/severe lung disorder requiring home-based oxygen therapy.
5. Patient requiring ECMO, hemodialysis or hemofiltration at the time of treatment administration.
6. Current diagnosis of pulmonary embolism.
7. Active neoplasm, except carcinoma in situ or basalioma.
8. Known allergy to the products involved in the allogenic MSC production process.
9. Current pregnancy or lactation (women with childbearing potential should have a negative pregnancy test result at the time of study enrollment).
10. Current participation in a clinical trial with an experimental treatment for COVID-19 (the use of any off-label medicine according to local treatment protocols is not an exclusion criteria).
11. Any circumstances that in the investigator's opinion compromises the patient's ability to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in the PaO2/FiO2* ratio from baseline to day 7 of treatment administration | 7 days
  Primary endpoint

SECONDARY OUTCOMES:
All-cause mortality | Days 7, 14, and 28 after treatment
  Secondary endpoint
Time to PaO2/FiO2 ratio greater than 200 mmHg | 12 months
  Secondary endpoint
Clinical status on the World Health Organization ordinal scale | Baseline, daily until day 14, and on day 28 after treatment
  Secondary endpoint.
  Categories:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  6. Hospitalized, on invasive mechanical ventilation or ECMO .
  7. Death.
PaO2/FiO2 ratio | Baseline and days 2, 4, 14 and 28 after treatment
  Secondary endpoint
SOFA score | Baseline and days 2, 4, 7, 14 and 28 after treatment
  Secondary endpoint Sequential Organ Failure Assessment score (0-24)
Oxygen therapy-free days | Day 28
  Secondary endpoint
Duration of hospitalization | 12 months
  Secondary endpoint
Duration of ICU admission | 12 months
  Secondary endpoint
Incidence of non-invasive ventilation | Day 28
  Secondary endpoint Proportion of patients with non-invasive ventilation
Incidence of invasive mechanical ventilation | Day 28
  Secondary endpoint Proportion of patients with invasive mechanical ventilation
Duration of non-invasive ventilation | Day 28
  Secondary endpoint (number of days)
Duration of invasive mechanical ventilation | Day 28
  Secondary endpoint (number of days)
Mechanical ventilation-free days | Day 28
  Secondary endpoint
Survival rate | 3 and 12 months.
  Secondary endpoint
Cumulative incidence SAEs, Grade 3 and 4 AEs, ADR and AEs of special interest. | 12 months
  Secondary endpoint

OTHER OUTCOMES:
Analytical endpoints | Baseline and days 2, 4, 7, 14 and 28 after treatment
  Exploratory endpoint Analytical markers (e.g., neutrophil and lymphocyte counts). Changes from baseline to set time points will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael F Duarte, MD, PhD, Study Chair — Hematology Department. Hospital Universitario Puerta de Hierro; Cristina Avedano-Sola, MD, PhD, Study Chair — Clinical Pharmacology Department. Hospital Universitario Puerta de Hierro; Juan J Rubio, MD, PhD, Principal Investigator — ICU. Hospital Universitario Puerta de Hierro; Rosa Malo, MD, Principal Investigator — Respiratory Medicine Department
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Munoz ME, Payares-Herrera C, Lipperheide I, Malo de Molina R, Salcedo I, Alonso R, Martin-Donaire T, Sanchez R, Zafra R, Garcia-Berciano M, Trisan-Alonso A, Perez-Torres M, Ramos-Martinez A, Ussetti P, Rubio JJ, Avendano-Sola C, Duarte RF. Mesenchymal stromal cell therapy for COVID-19 acute respiratory distress syndrome: a double-blind randomised controlled trial. Bone Marrow Transplant. 2024 Jun;59(6):777-784. doi: 10.1038/s41409-024-02230-5. Epub 2024 Feb 26. PMID 38409332
- [Derived] Payares-Herrera C, Martinez-Munoz ME, Vallhonrat IL, de Molina RM, Torres MP, Trisan A, de Diego IS, Alonso R, Zafra R, Donaire T, Sanchez R, Rubio JJ, Duarte Palomino RF, Sola CA. Double-blind, randomized, controlled, trial to assess the efficacy of allogenic mesenchymal stromal cells in patients with acute respiratory distress syndrome due to COVID-19 (COVID-AT): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Jan 6;22(1):9. doi: 10.1186/s13063-020-04964-1. PMID 33407777